CLINICAL TRIAL: NCT04225650
Title: Assessing the Prevalence of Respiratory Impairment in Chronic Inflammatory Bowel Diseases
Brief Title: Prevalence of Respiratory Impairment During IBD
Acronym: PARAMICI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: University of Lorraine (Other)
Responsible Party: Sponsor
Other Study IDs: 2019PI164
Record Dates: First submitted 2020-01-07; First posted 2020-01-13 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2019-12

CONDITIONS: Chronic Obstructive Pulmonary Disease; Asthma; Bronchiectasis; Inflammatory Bowel Diseases
Keywords: Chronic Obstructive Pulmonary Disease; Asthma; Epidemiology; Inflammatory Bowel Diseases
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Bronchiectasis; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pulmonology consultation — In case of functional respiratory signs, a consultation with a pulmonologist will be booked. At the end of this consultation, if the doctor deems it necessary, other investigations will be proposed and/or regular follow-up will be organised.

SUMMARY:
Patients will be recruited during a routine consultation with a physician in the hepato-gastroenterology department.

At the end of the consultation, patients will have to complete the following questionnaire: "European Community Respiratory Health Survey" which allows the screening of patients at risk of chronic respiratory diseases (asthma, COPD, bronchiectasis, emphysema).

In the event of a declaration of functional respiratory signs, a consultation with a pulmonologist will be systematically proposed. At the end of this consultation, if the doctor deems it necessary, further investigations will be proposed and/or regular follow-up organised.

The main objective of this study is to estimate the prevalence of respiratory symptoms leading to a diagnosis of chronic respiratory disease in patients with inflammatory bowel diseases (IBD) (Crohn's disease and UC).

The main criterion for judgement will be the frequency of functional respiratory signs (wheezing, dyspnea, cough, sputum) reported by IBD patients through an adapted self-report questionnaire.

DETAILED DESCRIPTION:
Approximately one-third of IBD patients will develop systemic extra-digestive manifestations (joint, dermatologic or ophthalmologic) during the course of their disease and up to 25% will develop these systemic manifestations even before the diagnosis of IBD. Among these systemic affections, respiratory manifestations remain poorly known because they are not searched for in daily clinical practice.

The main objective of this study is to estimate the prevalence of respiratory symptoms leading to a diagnosis of chronic respiratory disease (asthma, COPD, bronchiectasis) in patients with IBD (Crohn's disease and UC).

Patients will be recruited during a routine consultation with a physician in the hepato-gastroenterology department as part of the management of their chronic inflammatory bowel disease.

During this consultation, the investigating physician will explain to the patient the objective of the study and check with him/her the eligibility criteria. The patient will then be given an information note. He or she may ask any questions he or she wishes and if he or she refuses to participate in the study, he or she will have to sign an objection form in duplicate (one copy will be given to the patient and the other will be kept in the medical file). The doctor will also sign these two copies.

At the end of the consultation, patients will have to complete the following questionnaire: "European Community Respiratory Health Survey" which allows the screening of patients at risk of chronic respiratory diseases (asthma, COPD, bronchiectasis, emphysema).

In the event of a declaration of functional respiratory signs, a consultation with a pulmonologist from the Department of Pulmonology of the CHRU Nancy-Brabois will be systematically proposed. At the end of this consultation, if the doctor deems it necessary, further investigations will be proposed and/or regular follow-up organised. Patients will be informed of this potential follow-up in pneumology before the questionnaire is given. There is no change in the usual follow-up of the population in case of non-reporting of functional respiratory signs.

The main criterion for judgement will be the frequency of functional respiratory signs (wheezing, dyspnea, cough, sputum) reported by IBD patients through an adapted self-report questionnaire.

If our hypothesis is confirmed, this will have direct practical consequences on the global and multidisciplinary management of IBD patients, in particular through a systematic search for chronic respiratory disease, which is currently under-researched in these patients.

This will improve the quality of life as well as the morbidity and mortality of our patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with IBD (Crohn disease or Ulcerative colitis) between January 1990 and December 2019.
* Consultation in the Hepato-Gastroenterology Department of the CHRU Nancy-Brabois
* Patients who received full information about the research organization and did not object to the use of the data.
* Patients over 18 years of age

Exclusion Criteria:

* Inability to complete the questionnaire
* Diagnosis of IBD uncertain
* Persons referred to in Articles L. 1121-5, L. 1121-7 and L1121-8 of the Public Health Code :Pregnant, parturient or breastfeeding mother, Minor person, person who is subject to a legal protection measure
* Unable to express consent
* Persons deprived of their liberty by a judicial or administrative decision,
* Persons under psychiatric care (articles L. 3212-1 and L. 3213-1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult patient followed for IBD in the hepato-gastroenterology department of the CHRU de Nancy may be eligible.
Sampling Method: Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Frequency of functional respiratory signs | Through study completion, an average of 6 months
  Frequency of functional respiratory signs (wheezing, dyspnea, coughing, sputum) reported by IBD patients

SECONDARY OUTCOMES:
Chronic respiratory diseases | Through study completion, an average of 6 months
  Frequency of chronic respiratory diseases (asthma, COPD, respiratory allergies) among IBD patients
Exacerbations | Through study completion, an average of 6 months
  Frequency of reported exacerbations of chronic respiratory diseases in IBD patients.
Drugs | Through study completion, an average of 6 months
  Frequency of use of respiratory tropic drugs by IBD patients

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baumgart DC, Carding SR. Inflammatory bowel disease: cause and immunobiology. Lancet. 2007 May 12;369(9573):1627-40. doi: 10.1016/S0140-6736(07)60750-8. PMID 17499605
- [Background] Torres J, Mehandru S, Colombel JF, Peyrin-Biroulet L. Crohn's disease. Lancet. 2017 Apr 29;389(10080):1741-1755. doi: 10.1016/S0140-6736(16)31711-1. Epub 2016 Dec 1. PMID 27914655
- [Background] Ungaro R, Mehandru S, Allen PB, Peyrin-Biroulet L, Colombel JF. Ulcerative colitis. Lancet. 2017 Apr 29;389(10080):1756-1770. doi: 10.1016/S0140-6736(16)32126-2. Epub 2016 Dec 1. PMID 27914657
- [Background] Rodriguez-Roisin R, Bartolome SD, Huchon G, Krowka MJ. Inflammatory bowel diseases, chronic liver diseases and the lung. Eur Respir J. 2016 Feb;47(2):638-50. doi: 10.1183/13993003.00647-2015. Epub 2016 Jan 21. PMID 26797027